CLINICAL TRIAL: NCT02721459
Title: Phase I Study of Escalating Doses of XL888 With Vemurafenib Plus Cobimetinib for Patients With Unresectable BRAF Mutated Stage III/IV Melanoma
Brief Title: XL888 + Vemurafenib + Cobimetinib for Unresectable BRAF Mutated Stage III/IV Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Exelixis (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18597
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Skin Cancer
Keywords: unresectable melanoma; stage III melanoma; stage IV melanoma; AJCC melanoma staging; American Joint Committee on Cancer (AJCC); BRAF V600 E mutation; BRAF V600 K mutation
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Hsp90 inhibitor KU757; Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Escalating Doses of XL888 with Vemurafenib plus Cobimetinib.
  Interventions: Drug: XL888; Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: XL888 — Level 1: XL888 30 mg by mouth (PO) twice weekly (BIW). Level 2: XL888 45 mg PO BIW.
  Level 3: XL888 60 mg PO BIW. Level 4: XL888 90 mg PO BIW.
  Other Names: HSP90 inhibitor
Drug: Vemurafenib — Vemurafenib 720 mg by mouth twice a day (BID)
  Other Names: Zelboraf ®
Drug: Cobimetinib — Cobimetinib 40 mg by mouth once daily (QD). Administered 3 weeks on, 1 week off.
  Other Names: GDC-0973/XL518

SUMMARY:
The main purpose of this study is to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of XL888 when administered orally with vemurafenib plus cobimetinib in participants with BRAF V600 mutated melanoma and to evaluate the safety and tolerability of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or above. All races and ethnicities are eligible and no upper limit of age is specified.
* Must have cytologically or histologically-confirmed unresectable melanoma that harbors a BRAF V600 mutation determined by pyrosequencing assay or equivalent genotyping assay in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory, meeting one of the following AJCC staging criteria: 1.) American Joint Committee on Cancer (AJCC) stage IV (Tany, Nany, M1a, b, or c); 2.) AJCC stage IIIB or IIIC with unresectable nodal/locoregional involvement.
* Adequate hepatic, renal, and bone marrow function with parameters obtained within 4 weeks prior to initiation of study treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Willing to give written informed consent per institutional guidelines and must be able to adhere to dose and visit schedules.
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for ≥1 year.
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician.
* Treatment-naïve and previously treated patients will be included; however, patients may not have received a BRAF, Mitogen Activated Kinase (MEK) or HSP90 inhibitor in the past.
* May have received prior systemic and/or radiation therapy. All adverse events associated with prior systemic therapy or radiation therapy must have resolved to ≤ Grade 1 prior to start of study.
* Must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

Exclusion Criteria:

* Women who are pregnant, intend to become pregnant or are nursing.
* Previously treated with BRAF, MEK or HSP90 inhibitor therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy.
* Potential participants with untreated or uncontrolled brain metastases or evidence of leptomeningeal disease. Patients with asymptomatic brain metastases or previously treated brain metastases that are stable (i.e., not requiring corticosteroids) at the time of study start will be eligible.
* Previous malignancy is not an exclusion provided that the other malignancy is considered under control, patient is not on concomitant anti-cancer drug therapy, and target lesions from melanoma are clearly defined for response assessment.
* History of malabsorption or other condition that would interfere with absorption of study drugs.
* The following foods/supplements are prohibited at least 7 days prior to initiation of and during study treatment: St. John's wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer); Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor).
* Ocular: History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion (RVO), or neovascular macular degeneration.
* Cardiac: History of clinically significant cardiac dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 12 months
  The maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of XL888 when administered orally with vemurafenib plus cobimetinib in patients with BRAF V600 mutated melanoma.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/